CLINICAL TRIAL: NCT01402180
Title: A Randomized Phase II Trial Evaluating The Addition Of Nimotuzumab To Chemoradiation For Patients With Esophageal Squamous Cell Carcinoma After Radical Esophagectomy Who Suffer With Lymph Nodes Recurrence
Brief Title: Chemoradiation With or Without Nimotuzumab in Treating Esophageal Cancer Patients Who Suffer With Recurrence in Regional Lymph Nodes After Esophagectomy
Acronym: Nimotuzumab
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Xiao-Long Fu / Professor, Fudan University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010ESO_FU
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; lymph nodes recurrence; chemoradiation; Nimotuzumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients randomized in Arm A will receive chemoradiation and weekly Nimotuzumab for 6 weeks concurrent with radiation
  Interventions: Biological: Nimotuzumab; Radiation: Radiation therapy; Drug: chemotherapy
- B (Active Comparator): Patients randomized in Arm B will receive chemoradiation only
  Interventions: Radiation: radiation therapy; Drug: chemotherapy

INTERVENTIONS:
Biological: Nimotuzumab
  Arms: A
Radiation: Radiation therapy
  Arms: A
Radiation: radiation therapy
  Arms: B
Drug: chemotherapy
  Arms: A
Drug: chemotherapy
  Arms: B

SUMMARY:
A randomized phase II tials to study whether it's benefit of adding Nimotuzumab to chemoradiation for patients with esophageal squamous cell carcinoma after radical esophagectomy who suffer with locoregional lymph nodes recurrence.

DETAILED DESCRIPTION:
Patient population:

Esophageal squamous cell carcinoma after radical esophagectomy, then recurrent with lymph nodes in bilateral supravascular fossa or upper mediastinum 6 months beyond esophagectomy.

Scheme:

Eligible recurrent patients with esophageal cancer will first be stratified by recurrent time after esophagectomy (within 2 years after esophagectomy, or beyond 2 years after esophagectomy), then randomized to 2 arms at 1:1 ratio.

Arm A:

Chemoradiation + weekly Nimotuzumab for 6 weeks concurrent with radiation.

Arm B:

Chemoradiation only.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤75
2. ECOG performance status 0-2
3. Histologically proven primary thoracic esophageal squamous cell carcinoma before
4. Diagnosis of regional lymph nodes (biosupravascular fossa or upper mediastinum) recurrence after radical esophagectomy, based on pathological finding or imaging showing lymph nodes enlargement
5. Period from esophagectomy to diagnosis of regional lymph nodes recurrence should be more than 6 months
6. Without prior radiotherapy
7. Weight loss no more than 10% in the past 6 months
8. WBC≥ 4.0X109/L ,Absolute neutrophil count (ANC) ≥ 2.0X109/L
9. Platelets ≥ 100X109/L
10. Hemoglobin ≥ 90g/L(without blood transfusion)
11. AST (SGOT)/ALT (SGPT) ≤ 2.5 x upper limit of normal, Bilirubin ≤ 1.5 x upper limit of normal
12. Creatinine ≤ 1.5 x upper limit of normal
13. Sign study-specific informed consent prior to study entry

Exclusion Criteria:

1. With recurrence or metastasis other than regional lymph nodes (biosupravascular fossa or upper mediastinum)
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Severe, active comorbidity, defined as follows:

   3.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months 3.2 Transmural myocardial infarction within the last 6 months 3.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration 3.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration 3.5 Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
5. Prior radiation therapy or prior target drug therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Local control
  To evaluate if the addition of nimotuzumab to chemoradiation improves local control compared to chemoradiation only in patients with esophageal squamous cell carcinoma after radical esophagectomy who recurrent in regional lymph nodes.

SECONDARY OUTCOMES:
Overall survival
  To evaluate if the addition of nimotuzumab to chemoradiation improves overall survival compared to chemoradiation only in patients with esophageal squamous cell carcinoma after radical esophagectomy who recurrent in regional lymph nodes.
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Long Fu, M.D, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China